CLINICAL TRIAL: NCT02913794
Title: A Single-center Cross-sectional Study to Evaluate the Effectiveness of Antihypertensive Treatment Including Fimasartan and the Dyslipidemia Treatment Including Rosuvastatin and to Assess the Association Between the Two Treatments
Brief Title: Fimasartan and Rosuvastatin for Hypertension and Dyslipidemia Control
Acronym: FIMARO
Status: Completed | Type: Observational
Sponsor: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: BR-FMS-OS-402
Record Dates: First submitted 2016-09-21; First posted 2016-09-26 (Estimated); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Cardiovascular Diseases; Hyperlipidemias
MeSH Terms: conditions — Cardiovascular Diseases; Hyperlipidemias

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Fimasartan and Rosuvastatin for hypertension and dyslipidemia control

ELIGIBILITY:
Inclusion Criteria:

* Hypertension patients who are taking an anti-hypertensive agent, including Fimasartan at least 12 weeks or more.
* Dyslipidemia patients who are taking dyslipidemia drug, including Rosuvastatin at least 12 weeks or more
* Patients who has blood pressure and lipid levels (Total cholesterol, LDL-C, HDL-C, non-HDL-C, * TG) checks 2 weeks before registration

Exclusion Criteria:

* Patients being hospitalized
* Patients who stop taking Fimasartan or Rosuvastatin within 12 weeks 14 or more consecutive days
* Patients who have more than 400mg/dl triglyceride(TG) at the registration time

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1,056 patients
Sampling Method: Probability Sample
Enrollment: 541 (Actual)
Dates: Start 2016-10-11 (Actual); Primary Completion 2018-03-29 (Actual); Study Completion 2018-03-29 (Actual)

PRIMARY OUTCOMES:
Co-relation between blood pressure and dyslipidemia | 12 weeks
  Check the blood pressure and dyslipidemia control rates, also check the correlation between these two disease

CONTACTS AND LOCATIONS:
Overall Officials: Hyung-Jin Jung, Study Director — Boryung Pharmaceutical Co., Ltd
Locations (1):
- Severance Hospital, Seoul, South Korea